CLINICAL TRIAL: NCT00196066
Title: Evaluation of the Zilver Vascular Stent in the Iliac Arteries (ZIPS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 02-513
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Arterial Disease (PAD)
MeSH Terms: conditions — Peripheral Arterial Disease

INTERVENTIONS:
Device: Peripheral Vessel Stenting

SUMMARY:
The purpose of this study is to assess the ability of a vascular stent to maintain an open iliac (leg) artery. The Zilver Vascular Stent is made of nitinol, a flexible metal with a long history of use in medical devices. The stent self-expands once inside the artery where it is intended to hold the vessel wall open. Within a few weeks, a layer of cells will grow over the stent helping to hold it in place.

ELIGIBILITY:
Inclusion Criteria:

* Patient has documented stenotic or occluded atherosclerotic lesions of the external iliac or common iliac artery.
* Patient has a de novo or restenotic lesion(s) with no prior stent in the target lesion.
* Patient has given informed consent.

Exclusion Criteria:

* Patient is less than 50 years of age
* Patient is participating in another investigational drug or device study.
* Patient has multiple lesions (ipsilateral or in the aorta) that would require a staged procedure.
* Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* Patient has a known hypersensitivity or contraindication to aspirin, clopidogrel, nitinol, or contrast dye that cannot be adequately premedicated.
* Patient is pregnant or breast-feeding.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-10; Study Completion 2006-04

PRIMARY OUTCOMES:
The primary endpoint of the study is major adverse event (MAE) rate at the 9-month follow-up.

SECONDARY OUTCOMES:
Additional endpoints include acute procedure and hemodynamic success, secondary patency, 9-month restenosis rate based on ultrasound examination, and 9-month functional status improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Zemel, MD, Principal Investigator — Baptist Cardiac and Vascular Institute

REFERENCES:
- [Background] Krol KL, Saxon RR, Farhat N, Botti CF, Brown OW, Zemel G, Raabe RD, Voorhees WD 3rd, Katzen BT. Clinical evaluation of the Zilver vascular stent for symptomatic iliac artery disease. J Vasc Interv Radiol. 2008 Jan;19(1):15-22. doi: 10.1016/j.jvir.2007.08.031. PMID 18192463
- [Background] Jaff MR, Katzen BT. Two-year clinical evaluation of the Zilver vascular stent for symptomatic iliac artery disease. J Vasc Interv Radiol. 2010 Oct;21(10):1489-94. doi: 10.1016/j.jvir.2010.06.013. PMID 20801673